CLINICAL TRIAL: NCT01701180
Title: Neural Correlates of the Empathogenic and Affiliative Actions of Oxytocin
Brief Title: Neural Correlates of Empathogenic and Affiliative Actions of Oxytocin
Acronym: ODIS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, MSc MD PhD, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OXT-151/12; OXT-151/12 (Other Grant/Funding Number: HU1302/2-2 and NEMO)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Male Volunteers
MeSH Terms: interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): 24 IU Oxytocin, intranasal application 45 min prior to the experiment
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Intranasal application, sodium chloride solution, 3 puffs per nostril
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 24 IU; 3 puffs per nostril, each with 4 IU OXT
  Other Names: Oxytocin: Syntocinon-Spray, Novartis
  Arms: Oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Mounting evidence indicates that the intranasal administration of the neuropeptide oxytocin has prosocial effects. However, the neural substrates of these effects are still unclear. The investigators hypothesized that a single dose administration of oxytocin should increase empathogenic and affiliative responses and that these effects are mediated by an increased insula activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* In a heterosexual relationship

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Tobacco smokers

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Empathy ratings and their neural correlates | About one hour after the intranasal administration of oxytocin
  All subjects are scanned while they view emotional and neutral faces and rate their empathy for these stimuli.

SECONDARY OUTCOMES:
Neural correlates of pair-bonding | About one hour after the intranasal administration of oxytocin
  All subjects are scanned while they view a picture of their mate and and an unknown female.

CONTACTS AND LOCATIONS:
Overall Officials: René Hurlemann, MD PhD M.Sc., Principal Investigator — Department of Psychiatry University of Bonn
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- See also: NEMO research group — http://renehurlemann.squarespace.com/welcome/